CLINICAL TRIAL: NCT01292005
Title: Pentoxifylline Treatment in Acute Pancreatitis; A Double-Blind Placebo-Controlled Randomized Trial
Brief Title: Pentoxifylline Treatment of Acute Pancreatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Santhi Swaroop Vege, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-006648
Record Dates: First submitted 2010-10-19; First posted 2011-02-09 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-03

CONDITIONS: Acute Pancreatitis
Keywords: pancreatitis; pancreatic necrosis; severe acute pancreatitis (SAP); Alcoholic pancreatitis; gallstone pancreatitis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing; Pancreatitis, Alcoholic | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline (Experimental): Pentoxifylline, 400 mg, 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects received up to a maximum of 9 doses.
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Placebo, 400 mg, 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects received up to a maximum of 9 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — 400 mg, 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects received up to a maximum of 9 doses.
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — 400 mg, 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects received up to a maximum of 9 doses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects (good and bad) of giving a drug called pentoxifylline to patients with acute pancreatitis, to see if it can improve blood tests associated with inflammation (tissue damage). Pentoxifylline is approved by the US Food and Drug Administration (FDA) for treatment of circulation problems, but its use in this study is investigational, which means that the FDA has not approved it for the treatment of pancreatitis. However, the FDA has allowed the use of pentoxifylline in this research study.

DETAILED DESCRIPTION:
Subjects will be put in one of two groups by chance (as in the flip of a coin). This is done so that neither you nor the investigator will know which group you are in.

You will be put into either the treatment group or the control group.

* The treatment group will receive a drug called pentoxifylline
* The control group will receive a placebo (matching pill that has no medication in it) You will take the pills by mouth starting from the time of admission. You will receive a total of 9 doses over the first three days of your hospitalization (72 hours).

When subject have standard patient care blood draws, additional blood will be taken to do the research tests. The additional blood tests will be done every day for up to 5 days, after the administration of study drug or till the time of discharge whichever occurs earlier. The additional tests will require about 2 teaspoons (10 ml) of blood per day; the maximum amount of extra blood taken would be less than 3 tablespoons (40.0 ml). Information from your medical record will be gathered while you are hospitalized and after your discharge. The study will continue to gather clinical follow up information up to four months.

ELIGIBILITY:
Inclusion Criteria:

1. Predicted Severe Acute Pancreatitis
2. Enrollment within 72 hours of diagnosis
3. Ability to give informed consent
4. Age >17 years

Exclusion Criteria:

1. Moderate or severe congestive heart failure
2. History of seizure disorder or demyelinating disease
3. Nursing mothers
4. Pregnancy
5. History of prior tuberculosis or risk factors for tuberculosis
6. Evidence of immunosuppression (malignancy, chronic renal failure, chemotherapy within 60 days, ongoing steroid treatment*, and HIV)- (*the exception of prednisone use will be allowed to participate).
7. Evidence of chronic pancreatitis from history and examination (however, "acute on chronic pancreatitis" diagnosis is allowed)
8. Evidence of active or pending hemorrhage.
9. Paralytic ileus with vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santhi S Vege, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Vege SS, Atwal T, Bi Y, Chari ST, Clemens MA, Enders FT. Pentoxifylline Treatment in Severe Acute Pancreatitis: A Pilot, Double-Blind, Placebo-Controlled, Randomized Trial. Gastroenterology. 2015 Aug;149(2):318-20.e3. doi: 10.1053/j.gastro.2015.04.019. Epub 2015 Jun 23. PMID 26112745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from the Mayo Clinic in Rochester, Minnesota between 2009 and 2012.
Pre-assignment Details: 30 subjects signed informed consent; two subjects were excluded after consent because they were found to be not eligible.
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 69 [34 to 87] | 58 [24 to 82] | 64 [24 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Body Mass Index [Median (Full Range); unit: kg/m^2] | 30.2 [20.6 to 42.9] | 32.5 [16.7 to 50.1] | 30.3 [16.7 to 50.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in C-Reactive Protein (CRP)
Description: C-reactive protein is produced by the liver. The level of CRP rises when there is inflammation throughout the body. The normal value range for CRP = 1-10 mg/L.
Time Frame: baseline, Day 1, Day 3
Measure: Median (Full Range); unit: mg/L
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
mg/L
  Change from baseline to Day 1 | 48.4 [-37.1 to 207.3] | 60.6 [-71 to 283.2]
  Change from baseline to Day 3 | 62 [-157.4 to 255.3] | 154 [-170 to 193.5]
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 1. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 3. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 1.0, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Tumor Necrosis Factor (TNF)-Alpha
Description: Normal value range for TNF alpha = 0 - 22 pg/ml.
Time Frame: baseline, Day 1, Day 3
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
pg/ml
  Change from baseline to Day 1 | 0 [-1.2 to 0.52] | -0.05 [-0.9 to 49.2]
  Change from baseline to Day 3 | 0.2 [-1.0 to 0.5] | -0.3 [-3.5 to 17.2]
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 1. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 3. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Interleukin (IL) IL-6
Description: Normal value range for IL-6 = 0 - 5 pg/ml.
Time Frame: baseline, Day 1, Day 3
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
pg/ml
  Change from baseline to Day 1 | 2.1 [-37 to 25] | 0.7 [-62 to 152]
  Change from baseline to Day 2 | -8.6 [-61 to 15.6] | -2.9 [-213 to 65.8]
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 1. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.58, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 3. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Changes in Interleukin (IL) IL-8
Description: Normal value range for IL-8 = 0 - 5 pg/ml.
Time Frame: baseline, Day 1, Day 3
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
pg/ml
  Change from baseline to Day 1 | -3.0 [-7.2 to 30.8] | -1.7 [-38.2 to 49.2]
  Change from baseline to Day 3 | 0.35 [-10.3 to 5.4] | -1.9 [-43.6 to 18.2]
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 1. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Change from Day 0 to Day 3. p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number Of Subjects With New Onset Organ Failure During Hospitalization
Time Frame: 1 week or until dismissal date whichever occurs earlier.
Measure: Number; unit: participants
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
participants | 0 | 3
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number Of Subjects With New Onset Pancreatic Necrosis During Hospitalization
Time Frame: 1 week or until dismissal date whichever occurs earlier
Measure: Number; unit: participants
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
participants | 0 | 2
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; p<0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Patients With Lengthy Hospital Stays
Description: "Lengthy" was defined as either greater than 4 days or greater than 10 days.
Time Frame: 30 days or until dismissal date, whichever occurs earlier
Measure: Number; unit: participants
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
participants
  Length of hospitalization >4 days | 2 | 8
  Length of hospitalization >10 days | 0 | 5
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Comparison between arms for length of hospitalization > 4 days. P < 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.04, t-test, 2 sided
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Comparison was for length of hospitalization >10 days. P < 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

8. Secondary Outcome: Length of Hospital Stay
Time Frame: 30 days or until dismissal date, whichever occurs earlier
Measure: Median (Full Range); unit: days
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
days | 3 [1 to 5] | 5 [1 to 30]
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; P < 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

9. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Time Frame: 30 days or until dismissal date, whichever occurs earlier
Measure: Median (Full Range); unit: Days
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
Days | 0 [0 to 0] | 0 [0 to 13]
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; P < 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Subjects Who Needed an Intensive Care Unit Stay
Time Frame: 30 days, or until dismissal, whichever came first
Measure: Number; unit: participants
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 14 | 14
participants | 0 | 4
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; P < 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Pentoxifylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No